CLINICAL TRIAL: NCT01167816
Title: Phase I Trial of 5-Azacitidine Plus Gemcitabine in Patients With Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated as the Prinicipal Investigator left the site- all previous subjects enrolled are deceased
Sponsor: University of Oklahoma (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VZ-PANC-PI-0244
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- azacitabine (Experimental)
  Interventions: Drug: Vidaza

INTERVENTIONS:
Drug: Vidaza — Vidaza will be administered subq daily for 5 consecutive days each 28-day cycle
  Other Names: Azacitibine

SUMMARY:
The primary objective is to determine the maximum tolerated dose (MTD) of azacitidine and gemcitabine in subjects with previously untreated and unresectable pancreatic cancer. Also to determine the effect of azacitidine therapy on DNA methylation in peripheral blood cells.

DETAILED DESCRIPTION:
This is a Phase I single arm study designed for subjects with newly diagnosed, unresectable pancreatic cancer who have received no prior chemotherapy, radiation therapy, or surgery with curative intent for pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have pathologically confirmed diagnosis of pancreatic adenocarcinoma
* Must have measurable disease as defined by RECIST. RECIST evaluation must have occurred within 4 weeks prior to study entry
* Must have newly diagnosed, unresectable disease and have received no prior chemotherapy, radiation therapy or surgery with curative intent for pancreatic cancer
* Karnofsky performance status of greater than or equal to 70%
* Other significant medical conditions must be well controlled and stable in the opinion of the investigator for at least 30 days prior to Study Day 1
* Women of child bearing age must have negative serum pregnancy test prior to treatment

Exclusion Criteria:

* Known central nervous system tumor involvement
* Evidence of other active malignancy requiring treatment
* Clinically significant heart disease
* Active serious systemic disease, including active bacterial or fungal infection
* Active viral hepatitis or symptomatic HIV infection. Positive serology alone is not exclusionary
* Prior surgery with curative intent for pancreatic cancer
* Prior or current chemotherapy or radiation therapy for pancreatic cancer. Palliative radiation for distant metastases (excluding metastases in the abdominal region) is allowed
* Breast feeding, pregnant, or likely to become pregnant during the study
* known or suspected hypersensitivity to azacitidine or mannitol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose | 28 days
  There will be 5 planned cohorts that will receive the escalating doses of azicitidine and gemcitabine. There will be at least 3 patients in each cohort
Toxicity | 28 days
  To describe the toxicity associated with the use of this combination regimen

SECONDARY OUTCOMES:
Determine the effect of azacitidine therapy on DNA methylation in peripheral blood cells
  Perform multivariable regression models to explore and assess associations among changes in DNA methylation in peripheral blood cells, chemo effect on tumor (stable disease or shrinkage based on scans) and changes in tumor markers.

CONTACTS AND LOCATIONS:
Overall Officials: Osama Qubaiah, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Stephenson Cancer Center, Oklahoma City, Oklahoma, United States